CLINICAL TRIAL: NCT03767296
Title: Influence of a Bolus Administration of Ephedrine and Phenylephrine on the Spinal Oxygen Saturation, Measured With NIRS.
Acronym: NIRS BOLUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016/0644
Record Dates: First submitted 2017-05-10; First posted 2018-12-06 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Influence of Vasoactive Medication on Spinal Oxygenation
Keywords: spinal oxygenation; NIRS
MeSH Terms: interventions — Ephedrine; Phenylephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose Bolus of E-P-E (Experimental): Ephedrine Hydrochloride 3 MG/ML- Phenylephrine - Ephedrine Hydrochloride 3 MG/ML
  Interventions: Drug: Ephedrine Hydrochloride 3 MG/ML; Drug: Phenylephrine
- Dose Bolus P-E-P (Experimental): Phenylephrine- Ephedrine Hydrochloride 3 MG/ML - Phenylephrine
  Interventions: Drug: Ephedrine Hydrochloride 3 MG/ML; Drug: Phenylephrine
- Dose Bolus E-E-E (Experimental): Ephedrine Hydrochloride 3 MG/ML- Ephedrine Hydrochloride 3 MG/ML - Ephedrine Hydrochloride 3 MG/ML
  Interventions: Drug: Ephedrine Hydrochloride 3 MG/ML
- Dose Bolus P-P-P (Experimental): Phenylephrine-Phenylephrine-Phenylephrine
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Ephedrine Hydrochloride 3 MG/ML — Bolus group, according to the randomization. Multiple boluses with incremental doses might be needed, according to the MAP ('effect titration')
  Incremental doses if needed:
  Ephedrine (E): 6 mg, 6mg, 9 mg, 9 mg, 12 mg, …..(max 24mg/bolus) A total amount of 140 mg Ephedrine will not be exceeded.
  Titrated according to the desired effect (= MAP decrease < 20%)
  Arms: Dose Bolus E-E-E; Dose Bolus P-E-P; Dose Bolus of E-P-E
Drug: Phenylephrine — Bolus group, according to the randomization. Multiple boluses with incremental doses might be needed, according to the MAP ('effect titration')
  Incremental doses if needed:
  Phenylephrine (PE): 50μg, 50μg, 100μg, 100μg, 150μg, 150μg,…(max 500µg/bolus) A total amount of 1500 μg will not be exceeded. Titrated according to the desired effect (= MAP decrease < 20%)
  Arms: Dose Bolus P-E-P; Dose Bolus P-P-P; Dose Bolus of E-P-E

SUMMARY:
To evaluate the influence of vasoactive medication on the spinal vasculature, we have chosen patients scheduled for arterial dilation of the lower limb as our study population. In these patients the spinal cord perfusion is not compromised. However, most patients will suffer from hypotension during surgery, due to the non-invasive type of surgery and the vasodilating effects of the anesthetics. Therefore, bolus administration of vasoactive medication (ephedrine, phenylephrine) is routinely required in order to increase the blood pressure.

The aim of the study is to observe the influence of a bolus administration of ephedrine and phenylephrine on the spinal vasculature, measured by NIRS.

DETAILED DESCRIPTION:
During the preoperative visit, baseline MAP (mean arterial blood pressure) will be defined.

All patients receive standard anesthesia care during the surgical procedure. Before induction of anesthesia, 6 additional sensors (stickers) are applied to the back of the patient (at three levels: 2 at the upper thoracic level, 2 at the lower thoracic level and 2 at the lumbar region). 2 sensors are routinely applied to the forehead to measure the cerebral oxygenation and a BIS sensor is applied to measure the depth of anesthesia. Through an intravenous line anesthetics will be administered. Vasopressor agents will be administered through a second intravenous line. After induction of anesthesia, an endotracheal tube is placed. According to the estimated duration of surgery a bladder catheter is placed.

If - after induction of anesthesia- MAP has decreased more than 20%, a vasopressor agent will be administered in order to increase the blood pressure to normal (preoperative) values. According to the MAP, several bolus administrations and incremental bolus dosages might be needed to reach the target blood pressure range (MAP decrease less than 20%). According to the group to which the patient has been randomized, a bolus of ephedrine and/or phenylephrine will be administered.

The study will be completed when MAP decreases more than 20% from baseline for the 4th time.

A total amount of Ephedrine and Phenylephrine resp. of 140 mg and 1500 μg will not be exceeded.

If the administration of the vasopressor study medication does not achieve the desired result, the patient will receive an appropriate treatment.

The endovascular surgical procedure can start without delay and the duration of surgery will not be prolonged because of the measurements and blood pressure management.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18y
* scheduled for dilation of arterial blood vessels of the lower limb

Exclusion Criteria:

* Age < 18y
* BMI > 30
* severe valvular disease
* previous aortic surgery
* paraplegia/ paraparesis
* renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-09-09 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
Spinal oxygen saturation measured by NIRS | from first till 4th MAP decrease > 20 % from baseline
  Spinal oxygen saturation measured by NIRS

SECONDARY OUTCOMES:
Heart rate | from first till 4th MAP decrease > 20 % from baseline
  Heart rate
Blood pressure | from first till 4th MAP decrease > 20 % from baseline
  Blood pressure
Cerebral oxygenation (NIRS) | from first till 4th MAP decrease > 20 % from baseline
  Cerebral oxygenation (NIRS)
Total amount of vasoactive medication used | from first till 4th MAP decrease > 20 % from baseline
  Total amount of vasoactive medication used

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Vanpeteghem, Principal Investigator — UZ Ghent
Locations (1):
- University Hospital Ghent, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vanpeteghem CM, Bruneel BY, Lecoutere IM, De Hert SG, Moerman AT. Ephedrine and phenylephrine induce opposite changes in cerebral and paraspinal tissue oxygen saturation, measured with near-infrared spectroscopy: a randomized controlled trial. J Clin Monit Comput. 2020 Apr;34(2):253-259. doi: 10.1007/s10877-019-00328-6. Epub 2019 Jun 5. PMID 31165350